CLINICAL TRIAL: NCT04473313
Title: Educational Follow-up in COPD Patients After Pulmonary Rehabilitation: a Cohort Study
Brief Title: Educational Follow-up in COPD Patients After Pulmonary Rehabilitation.
Acronym: EDURESPI
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0212 - EDURESPI
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After pulmonary rehabilitation, the challenge is to maintain the benefits reached during the program and increase physical activity.

As exercise training, education is the corner stone of pulmonary rehabilitation. Education allows to support behavioral changes in daily life.

Recommendations about modalities for maintaining physical activity are still clear, however for educational follow up recommendations need to be clarified.

After a pulmonary rehabilitation program, there is no defined plan for educational follow up nor location to perform education session.

The aim of this study is to evaluate the proportion of patients who succeed to establish and maintain the objectives they defined during the pulmonary rehabilitation program, one year after this program.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients COPD patients admitted for pulmonary rehabilitation program in pulmonary rehabilitation unit of CH des Pays de Morlaix or CHU Brest

Exclusion Criteria:

* inability to answer to the questionnaire
* refusal to participate.
* inability to perform the pulmonary rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients, all stages
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Realization of the objective(s) defined by the patient during a common educational assessment (educational diagnosis) at the end end of the pulmonary rehabilitation program | one year
  Determination of the objective(s) defined by the patient during a common educational assessment (educational diagnosis) at the end of the pulmonary rehabilitation program and evaluation of the realization of this (these) objective(s) after one year (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Beaumont, PhD, Principal Investigator — CH des pays de Morlaix
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - BEAUMONT, Morlaix

REFERENCES:
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Peran L, Le Ber C, Pichon R, Cabillic M, Beaumont M. [Follow-up and evaluation of plans developed during pulmonary rehabilitation]. Rev Mal Respir. 2018 Nov;35(9):929-938. doi: 10.1016/j.rmr.2018.08.002. Epub 2018 Sep 7. French. PMID 30201399